CLINICAL TRIAL: NCT04873076
Title: Change of Analgosedation (Remifentanil) Dosage and Increased Patient Satisfaction During Catheter Ablation Procedures in Cardiac Rhythm Disorders Via 2d Audiovisual Distraction.
Brief Title: Audiovisuell Distraction Via 2d Videoglasses During Catheter Ablation Procedures in Cardiac Rhythm Disorders.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-8325-BO
Record Dates: First submitted 2020-01-25; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Rhythm; Disorder
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audiovisual distraction using 2d video glasses from HappyMed GmbH (Experimental): During the catheter ablation, the patients in the intervention group receive 2D video glasses with headphones. Immediately before and after the procedure they receive a questionnaire. During the procedure vital parameters of all patients regardless of the studygroup are monitored using "Zoll X-Series Monitor Defibrillator. The study includes blood pressure (in mmHg), heart rate (in beats per minute) and patient's level of alertness, which is assessed using the Richmond Agitation-Sedation Scale(RAAS). During the procedure the patients in the intervention group receive the glasses and remote control. All patients receive their individual dosage to ensure painless ablation. The drugs used are limited to the opioids remifentanil and benzodiazepine midazolam.
  Interventions: Device: Audiovisual distraction using 2d video glasses from HappyMed GmbH
- Controll arm (No Intervention): In patients in the control group, catheter ablation is performed as usual without the use of video glasses. They receive immediately before and after the ablation the same questionnaire as the patients in experimental arm. (Omitting the question about the videoglasses).
  While the procedure is performed, the analgosediation is as well in the controll arm as in the experimental arm titrated until the patient is treated, sedated and painless.

INTERVENTIONS:
Device: Audiovisual distraction using 2d video glasses from HappyMed GmbH — Patients receive optical and acustical relaxing material during the procedure by using 2d video glasses from HappyMed GmbH
  Arms: Audiovisual distraction using 2d video glasses from HappyMed GmbH

SUMMARY:
In this randomized controlled trial, amount of sedation exposure and patient satisfaction is evaluated in patients undergoing catheter ablation for rhythm disorders via an audiovisual distraction. Patients are randomized into intervention group (adiovisual distraction) or controll (no intervention).

DETAILED DESCRIPTION:
Study conduct:

After the patient has been informed and given written consent to participate in the study, the patients are randomized. They are either assigned to the control group (in which catheter ablation will take place without video glasses as before) or to the intervention group in which they receive the video glasses during ablation. The randomization into the two groups is done by random allocation.

The patients in the intervention group receive instruction on how to use the video glasses and can familiarize themselves with them. Before the patient (as well in the intervention as in the control group) is taken to the EPU laboratory, he receives the first questionnaire in which the personal data and his mood / feeling of fear are collected. In addition, two questions on instrumental-qualification media studies should give an indication of possible relationships between the evaluation of video glasses. The patient is then led into the laboratory and connected to the monitoring by the team. Before it is covered under sterile conditions, the patients in the intervention group receive the glasses and remote control with which they can select the footage from the media library.

The anesthetist will inject a basic dose of sedative and analgesic (determined on the basis of body weight) into each patient and increase it if pain or agitation is noticeable. All patients receive their individual dosage to ensure painless ablation. During the examination, the vital parameters (blood pressure and heart rate) are documented at specified times.

After completing catheter ablation, the video glasses (for patients from the intervention group) are removed. The patients receive a second questionnaire in which they evaluate the use of the video glasses.

Both the subjects in the intervention and control groups are asked to estimate the duration of the examination. The subjective sense of time is intended to provide information as to whether the patients in the intervention group experienced adequate distraction compared to the patients in the control group.

Follow-up:

On the day after catheter ablation all patients receive the CSQ 8 questionnaire, which assesses patient satisfaction using categorical questions. A longer-term follow-up is not necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing catheter ablation for rhythm disorders

Exclusion Criteria:

* epilepsy
* age <18 years
* visus <-5 dpt or >+2 dpt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Change of analgosedation dosage | during the procedure (electrophysiological examination on the heart)
  The change of analgosedation dose is measured by comparing the amount of sedation necessary for the procedure in experimental and controll arm.
  Remifentanyl (Ultiva) is measured in µg/kg/hour Midazolam (Dormicum) is measured in mg/kg/hour
Change of stress and anxiety level | during the procedure (electrophysiological examination on the heart)
  The vital parameter blood pressure (in mmHg) serve as surrogate parameter for anxiety and stress.

SECONDARY OUTCOMES:
Patient satisfaction | evaluation before, immediately after and one day after the procedure
  Patient satisfaction is assessed using the established Client Satisfaction Questionnaire (CSQ-8). It consists of eight items on ordinal scale level. Each question has formulated answer options that correspond to a value from 1 to 4 with higher scores indicating higher satisfaction. The total score can range from 8 to 32.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No